CLINICAL TRIAL: NCT02286492
Title: An Open-Label Expanded Access Study of TAS-102 in Patients With Metastatic Colorectal Cancer Refractory to or Failing Standard Chemotherapy
Brief Title: Expanded Access Study of TAS-102 in Patients With Metastatic Colorectal Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TO-TAS-102-401
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — trifluridine tipiracil drug combination

INTERVENTIONS:
Drug: TAS-102 — At a dose of 35 mg/m2 administered orally twice daily for 5 days a week with 2 days rest for 14 days, followed by a 14-day rest (1 treatment cycle)

SUMMARY:
The objective of the program is to provide access to TAS-102 to patients with metastatic colorectal cancer who are refractory to or failing standard chemotherapy, are new to therapy with TAS-102 and in whom therapy with TAS-102 is clinically indicated.

DETAILED DESCRIPTION:
This is an open-label study to provide expanded access to TAS-102 prior to its commercial availability for patients with metastatic colorectal cancer who have been previously treated with, or are not candidates for fluoropyrimidine-, irinotecan-, and oxaliplatin-based chemotherapy, an anti-vascular endothelial growth factor (VEGF) therapy, and an anti-epidermal growth factor receptor (EGFR) therapy.

Serious adverse event information (whether or not related to TAS-102) as well as reports of pregnancy, overdose, or medication error will reported. In addition, all grades of adverse drug reactions (ADRs, adverse events related to study medication) and any adverse event that results in treatment discontinuation will be recorded as study data on CRFs.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has adenocarcinoma of the colon or rectum
3. Has failed at least 2 prior regimens of standard chemotherapies for metastatic colorectal cancer
4. ECOG performance status of 0 or 1
5. Is able to take medications orally
6. Has adequate organ function (bone marrow, kidney and liver)
7. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Certain serious illnesses or medical condition(s)
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, within the specified time frames prior to study drug administration
3. Has received TAS-102
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Alabama Oncology, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Global Cancer Research Institute (GCRI), Inc., Gilroy, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Pacific Hematology Oncology Associates (PHOA), San Francisco, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Florida Health Davis Cancer Center, Gainesville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Rochester, Rochester, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Dunmore, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fox Valley Hematology & Oncology, Appleton, Wisconsin

REFERENCES:
- [Derived] Mayer RJ, Hochster HS, Cohen SJ, Winkler R, Makris L, Grothey A. Safety of trifluridine/tipiracil in an open-label expanded-access program in elderly and younger patients with metastatic colorectal cancer. Cancer Chemother Pharmacol. 2018 Dec;82(6):961-969. doi: 10.1007/s00280-018-3686-5. Epub 2018 Oct 22. PMID 30350179